CLINICAL TRIAL: NCT07153185
Title: A Retrospective Multi-center, PMCF Study to Assess the Safety and Performance of a Biodegradable Dental Barrier Membrane (Creos Xenoprotect)
Brief Title: Creos Xenoprotect PMCF
Status: Not yet recruiting | Type: Observational
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Other Study IDs: T-195
Record Dates: First submitted 2025-08-15; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Bone Regeneration; Dental Implants; Bone Grafting
Keywords: Dental Barrier Membrane; PMCF Study; Retrospective

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- main study population
  Interventions: Device: Dental Barrier Membrane

INTERVENTIONS:
Device: Dental Barrier Membrane — Patients treated with creos xenoprotect dental barrier membrane in the past

SUMMARY:
The goal of this retrospective PMCF study is to assess safety and performance of creos xenoprotect in all indications functioning as dental barrier membrane.

The primary endpoint of the study is the occurrence of major complications during 6 months after creos xenoprotect placement whereas the hypothesis is that these major complications occur in less than 5% within this timeframe.

This is a retrospective, multicenter clinical investigation with consecutive cases. Data will be collected on consecutive data cases from patient files, given that these patients were treated within a defined indication with creos xenoprotect in the past. Patients participating in this study do not have any obligations or need to come back for any intervention. A total of 11 centers are planned to be included. Sample size is n=200 patients and is distributed equally in four indication groups:

Group 1: Ridge augmentation (vertical and horizontal) Group 2: Alveolar ridge preservation Group 3: Sinus floor augmentation Group 4: Augmentation around implant or teeth

ELIGIBILITY:
Inclusion Criteria:

* Participant was treated before December 2023 (creos xenoprotect placement)

  * Participant signed informed consent form and data protection consent form1
  * Participant was at least 18 years old at the time of treatment
  * Participant received guided bone regeneration combined with the use of creos xenoprotect according to one of the four indications
  * Participant was treated according to instructions for use (IFU)
  * Participant should have follow-up time of >9 months after placement of the investigational device

Exclusion Criteria:

* In Group 3: Sinus floor augmentation (lateral approach): usage of creos xenoprotect to replace a ruptured Schneiderian Membrane

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants (aged ≥ 18y) that underwent guided bone regeneration combined with the use of creos xenoprotect according to one of the four indications are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major complications during 6 months after creos xenoprotect placement | From Surgery to 6 Months Follow-Up

SECONDARY OUTCOMES:
Occurence of minor complications (dehiscence, membrane exposure, infection) during 6 months after placement of creos xenoprotect | From Surgery to 6 Months Follow-Up
Number of cases with successful bone graft: o Implants: sufficient bone at implant insertion visit o No implants: additional bone grafting intervention needed at 6 Months Follow-Up | From Surgery to 6 Months Follow-Up
Clinician satisfaction / handling with creos xenoprotect at Membrane Placement (VAS Scale) | At Surgery
  Visual Analog Scale, Score 1-10, 1: not satisfied at all; 10: totally satisfied
SAE, SADE, USADE, DD | From Surgery to 9 Months Follow-Up

OTHER OUTCOMES:
Implant survival (at final prosthesis delivery and last follow-up) | From Surgery to 9 Months Follow-Up
Bone gain (between membrane placement and follow-up visits) | From Surgery to 9 Months Follow-Up
Bleeding Index | From Final Prosthesis Placement to 9 Months Follow-Up
Plaque Index | From Final Prosthesis Placement to 9 Months Follow-Up
Gingival Index | From Final Prosthesis Placement to 9 Months Follow-Up
Keratinized Mucosa Height | From Final Prosthesis Placement to 9 Months Follow-Up
  [mm]
Gingival Thickness | From Final Prosthesis Placement to 9 Months Follow-Up
  [mm]
Buccal Soft Tissue Thickness | From Final Prosthesis Placement to 9 Months Follow-Up
  [mm]